CLINICAL TRIAL: NCT00918593
Title: Palliative Treatment of Ulcerated Cutaneous Metastases: Randomised Trial Between Electrochemotherapy and Radiotherapy
Brief Title: Palliative Treatment of Ulcerated Cutaneous Metastases: Trial Between Electrochemotherapy and Radiotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment of patients
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA0906; EudraCT number: 2009-011455-51
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Ulcerated Cutaneous Metastases
Keywords: Metastases; Cutaneous; Ulcerating; Palliative; ulcerating metastases
MeSH Terms: conditions — Neoplasm Metastasis; Ulcer | interventions — Electrochemotherapy; Radiotherapy; Bleomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrochemotherapy (Experimental)
  Interventions: Drug: Electrochemotherapy; Drug: Bleomycin
- radiotherapy (Active Comparator)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Drug: Electrochemotherapy — Intratumoral or intravenous bleomycin followed by electric pulses. Once only treatment.
  Other Names: ECT
  Arms: Electrochemotherapy
Radiation: Radiotherapy — Radiotherapy according to hospital procedures.
  Other Names: RT
  Arms: radiotherapy
Drug: Bleomycin — Intratumoral or intravenous bleomycin followed by electric pulses. Once only treatment.
  Arms: Electrochemotherapy

SUMMARY:
By applying short electric pulses to cells, the cell membranes can become permeabilised (electroporation). This can be used augment the effect of chemotherapy, by providing direct access to the cell cytosol. For the drug bleomycin, the enhancement of effect is several hundred fold, enabling once-only treatment. The investigators wish compare electrochemotherapy with radiotherapy when treating ulcerated cutaneous metastases up to 5 cm in diameter from any kind of histology.

DETAILED DESCRIPTION:
About 5 % of all cancer patients experience cutaneous metastases. Ulcerating metastases can be of great psychological distress for the patients and may also be painful. Radiation therapy is standard treatment for ulcerating metastases, but there are no reports of response rate.

With this study we wish to compare electrochemotherapy with radiotherapy when treating ulcerated cutaneous metastases up to 5 cm in diameter from any kind of histology.

Patient recruitment: 98 patients are to be recruited, the patients will be randomized between electrochemothreapy or radiotherapy. 49 patients will be treated in each arm.

Treatment: Patients will be treated in local or general anesthesia (inhaling max. 30 % oxygen) Bleomycin will be given either intratumoral or intravenous. Electric pulses will be administered using a square wave electroporator (IGEA, Carpi, Italy). Needle and plate electrodes are used in order to treat the affected area efficiently. Eight pulses at a frequency of 5000 Hz or 1 Hz will be used for each application of the electrodes. In this way, a large area can be treated within a short time. Post treatment, the area will be covered by dry dressings, as are standardly used.

The patients will be seen at 8, 30, 60, 90 and 180 days post treatment. Chest X ray will be taken before and after treatment for the patients receiving electrochemotherapy.

Evaluation: Evaluation is performed by measurement of lesion extension and digital photography using the RECIST criteria. The first 10 patients in each treatment arm will also be PET/CT-scanned before and one week after treatment.

Safety: Safety will be reported both in terms of evaluation of adverse events and in terms of patient satisfaction determined by questionnaire, including the 'Derriford Appearance Questionaire'.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18.
* Histological proven cancer, any histology.
* Progressive and/or metastatic disease.
* One or more ulcerating cutaneous metastases.
* Patient in need of palliation of the ulcerating metastases.
* Lesion to be treated between 1 cm - 5 cm in diameter.
* Lesions to be treated must be either stationary or progressing during any concomitant chemotherapy.
* WHO performance ≤ 2.
* Life expectancy of at least 3 months.
* Platelets ≥ 50 mia/l, pp ≥ 40, APTT in normal area. Medical correction is allowed.
* Sexual active men and women must use safe anticonceptive during and up to 6 month after last treatment.
* Written informed consent must be obtained according to the local Ethics committee requirements.

Exclusion Criteria:

* Previous electrochemotherapy or radiotherapy in the area to be treated
* Acute lung infection
* Previous bleomycin treatment exceeding 200.000 Units/m2.
* Known hypersensitivity to any of the components of the treatment.
* Known hypersensitivity to any of the components used in the planned anaesthesia.
* Pregnant or lactating women. In fertile women this is ensured by measuring HCG in blood.
* Treatment with granulocyte colony stimulating factor (G-CSF) or other cytokines.
* Creatinine measurements over 150 micromolar will require Crohm-EDTA clearance. Crohm-EDTA below 48 ml/minute
* Abnormal DLCO. If clinical history of or suspected reduced lung capacity, DLCO must be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2009-12; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Safety and response | 30 days

SECONDARY OUTCOMES:
patient satisfaction | 180
Economics | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, Consultant, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital at Herlev, Herlev, Copenhagen, Denmark